CLINICAL TRIAL: NCT03742310
Title: Multi-Center Clinical Study on the Relationship Between Vitamin D Receptor Gene Polymorphism and Children's Physical and Intellectual Development
Brief Title: The Relationship Between VDR Gene Polymorphism and Children's Physical and Intellectual Development
Acronym: RVDRGPCPID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xian Children's Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX201856
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-07

CONDITIONS: Development, Child
Keywords: Vitamin D Receptor gene; physical development; intelligent development
MeSH Terms: interventions — Vitamin D; Calcitriol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- identical supplement group (Experimental): Take vitamin D supplements according to genotype. If the genotype result is "high risk", we will give vitamin d 800 international unit(IU)/d, when the result is "middle risk", we will give 600 international unit(IU)/d, when the result is "low risk", we will give 400 international unit(IU)/d.
  Interventions: Drug: Vitamin D
- control group (No Intervention): General dose. Whatever the result is, we all give 400 international unit(IU)/d.

INTERVENTIONS:
Drug: Vitamin D — Vitamin D is essential for healthy bones, and to control the amount of calcium in our blood.It is important at every stage of life, but especially for rapidly growing infants and teenagers and for pregnant and breastfeeding women.
  Other Names: calcitriol
  Arms: identical supplement group

SUMMARY:
This study was used to determine the relationship between vitamin D receptor gene polymorphism and children's physical and intellectual development, further adjust the doses of vitamin D supplementation after birth, and provide individualized vitamin D and calcium supplements.

DETAILED DESCRIPTION:
High risk children aged 0-3 years old who visited the pediatrics clinic and ward of the first affiliated hospital of Xi'an Jiaotong university and other cooperative hospitals from 2018 to 2020 were randomly selected. Personal information of the children and parents who were enrollment was collected by questionnaire survey and a follow-up file was established. 500 to 1,000 people are planned to participate in the study, were randomly divided into research group and the control group. Then collect the sample(saliva) of children to examine Vitamin D Receptor(VDR) genotype, according to results, divide the research group into high, medium and low risk, given individual vitamin D and calcium supplement. Monitor the children's weight, body length, head circumference, the Neonatal Behavioral Assessment Scale(NBAS), bailey rating scale respectively, up to 3 years old. All sample analyses were performed by the Gene Medical Laboratory. Laboratory personnel were blinded to mother and infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* infant age from 0 to 3 years old
* enjoy good health, there is no history of specific diseases

Exclusion Criteria:

* this time or always exists serious lung infection, or with nervous system disease, kidney disease, malignant tumor, etc
* has bone metabolic diseases or other genetic metabolic disease
* taking affect bone metabolism of drugs for a long time

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
body weight | From date of randomization until the date of three year-old
  We will use the baby scale to measure infant body weight
body height | From date of randomization until the date of three year-old
  We will use the baby scale to measure infant body height
head circumference | From date of randomization until the date of three year-old
  We will use the tape to measure infant head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Hui Li, PHD,MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided